CLINICAL TRIAL: NCT05139394
Title: Emergency Pancreaticoduodenectomy: a Non-trauma Center Case Series
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Diana Schlanger, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: EPD - CS
Record Dates: First submitted 2021-09-29; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Emergencies; Pancreas Disease
MeSH Terms: conditions — Emergencies; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: emergency pancreaticoduodenectomy — Emergency pancreaticoduodenectomy (EPD) is a complex surgical procedure, that can be performed for complex pancreaticoduodenal injuries, that cannot be controlled through less invasive procedures. EPD can be performed either as a classical Whipple procedure, or as a pylorus-preserving procedure. A one stage procedure implies the reconstruction step being done in the same surgical intervention, while a two step procedure implies the reconstruction being done in a later stage, through a second surgical intervention.

SUMMARY:
Pancreaticoduodenectomy is a challenging procedure itself, being even more complex and demanding in emergency settings. Only a few cases of emergency pancreaticoduodenectomy (EPD) are reported in medical literature, usually performed for complex pancreaticoduodenal lesions. EPD has first been mentioned in trauma settings, even fewer cases being reported for non-traumatic indications. The investigators intend to present our experience with this intervention, in a non-trauma surgical centre. Our study is a prospective consecutive case series, that included patients that underwent emergency pancreaticoduodenectomy from January 2014 to May 2021. Data was collected from the electronic system database. The investigators collected data regarding the demographic characteristics of the patients, their medical history, preoperative and postoperative investigations (including blood work and imagistic investigations), surgery related information and postoperative evolution.

ELIGIBILITY:
Inclusion Criteria:

* Emergency pancreaticoduodenectomy performed

Exclusion Criteria:

* Elective surgery
* Insufficient data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated in Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor Cluj-Napoca January 2014 and May 2021
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | The length of the surgical intervention (an average of 3 hours)
  ml of blood
Operative time | The length of the surgical intervention (an average of 3 hours)
  minutes of operating time
In-hospital Morbidity | Up to 90 days. Through study completion, during the hospital admission period
In-hospital Mortality | Up to 90 days. Through study completion, during the hospital admission period
Long-term evolution | The date of the last follow-up information was August 2021
  It will be measured the overall survival time, number of readmissions and number of reinterventions

IPD SHARING:
Plan to Share IPD: Undecided